CLINICAL TRIAL: NCT01735877
Title: Effectiveness of Mirror Therapy in Stroke Patients With Unilateral Neglect - A Randomized Controlled Trial
Acronym: MUST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Responsible Party: Principal Investigator, jeyarajpandian, Professor, Christian Medical College and Hospital, Ludhiana, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MT2012
Record Dates: First submitted 2012-11-26; First posted 2012-11-28 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-05

CONDITIONS: Hemispatial Neglect
Keywords: Hemispatial neglect, Stroke
MeSH Terms: conditions — Perceptual Disorders; Stroke | interventions — Mirror Movement Therapy; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror therapy (Experimental): All eligible patients will be randomly allocated into 2 groups. Group 1 will be given Mirror therapy
  Interventions: Other: Mirror therapy
- Control group (Sham Comparator): Group 2 will be given sham mirror therapy
  Interventions: Other: Control group

INTERVENTIONS:
Other: Mirror therapy — During the mirror practices, patients were seated close to a table on which a mirror (35×35cm) was placed vertically. The practice consisted of non paretic-side wrist and finger flexion and extension movements while patients looked into the mirror, watching the image of their noninvolved hand, thus seeing the reflection of the hand movement projected over the involved hand. Patients could see only the noninvolved hand in the mirror; otherwise, the noninvolved hand was hidden from sight. During the session patients were asked to try to do the same movements with the paretic hand while they were moving the non paretic hand.
  Arms: Mirror therapy
Other: Control group — The control group performed the same exercises for the same duration but used the nonreflecting side of the mirror in such a way that the paretic hand was hidden from sight. The same therapist delivered the control therapy to the patients. Both the treatment and the control group received limb activation.
  Arms: Control group

SUMMARY:
Hemi spatial neglect, or the tendency to ignore stimuli originating in a portion of the environment contra lateral to a cerebral lesion, can be a major source of functional handicap after stroke. The currently available treatments for unilateral neglect are scanning training, visual cuing approaches, limb activation strategies, visual imagery, tactile stimulation, prisms and sustained attention training.Mirror therapy improves the hand function in sub-acute stroke.

Hypothesis: To evaluate the effectiveness of Mirror therapy in the management of stroke patients with unilateral neglect.

DETAILED DESCRIPTION:
About 30 - 50% of stroke patients are left with considerable residual deficits. The post stroke disabilities are due to loss of locomotion and activities of daily living, cognition and communication skills.Hemispatial neglect has been reported in association with damage to several different cerebral structures in a large-scale distributed neurocognitive network.Mirror therapy improves the hand function in sub-acute stroke. It also helps in the recovery of neglect in stroke patients. But little consensus exists as to whether one treatment is more efficacious than others and many studies fail to document duration of treatment effects or generalization to daily activities. The aim of our study is to evaluate the effectiveness of limb activation with MT and limb activation strategy alone in the management of stroke patients with unilateral neglect and to make the patient functional in activities of daily living.

ELIGIBILITY:
Inclusion Criteria: 1.All stroke patients with parietal lobe and thalamic lesions 2. Stroke duration: within 48 hours 3. Patients willing to participate in the study 4. MRI/ CT scan showing parietal lobe and thalamic lesion 5. Patients with upper limb weakness

Exclusion Criteria:

1. Stroke duration more than 1 yr
2. Glasgow Coma Scale (GCS) of less than 7
3. Uncooperative patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeyaraj Pandian, DM, Principal Investigator — BFUHS
Locations (1):
- Department of Neurology, CMC &H, Ludhiana, Punjab, India

REFERENCES:
- [Derived] Pandian JD, Arora R, Kaur P, Sharma D, Vishwambaran DK, Arima H. Mirror therapy in unilateral neglect after stroke (MUST trial): a randomized controlled trial. Neurology. 2014 Sep 9;83(11):1012-7. doi: 10.1212/WNL.0000000000000773. Epub 2014 Aug 8. PMID 25107877

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: January 2011 to August 2013
Period: Overall Study
Arm/Group | Mirror Therapy | Control Group
Started | 27 | 21
Completed | 26 | 21
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirror Therapy | Control Group | Total
Number analyzed (Participants) | 27 | 21 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.15 (11.07) | 64.29 (12.02) | 63.65 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  India | 27 | 21 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Star Cancellation Test Scores at 1,3, and 6 Months
Description: The SCT consisted of a page containing 52 large stars, 10 short words and 13 letters, randomly positioned, with 56 small stars interspersed. Subjects were instructed to cross out (with a black pen) all the small stars across the page. The tester demonstrated by crossing out the two central stars. The cut off score to establish presence of unilateral visual neglect were: 51 or fewer stars cancelled for SCT.
  Minimum score: 0 Maximum score: 54
  Higher scores: better outcome
Time Frame: Baseline, 1,3 and 6 months
Population: The number of participants are different as mentioned in the flow algorithm since 1 patient from the control group died at 3 months follow up. This patient is included in secondary outcome measures i.e. modified Rankin Scale (mRS)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mirror Therapy | Control Group
Number analyzed (Participants) | 26 | 20
units on a scale
  Baseline | 17.88 [15.91 to 19.85] | 18.20 [15.58 to 20.82]
  Baseline to 1 month | 20.03 (4.71) [17.98 to 22.09] | 5.90 (5.60) [3.55 to 8.24]
  Baseline to 3 month | 31.76 (5.19) [29.18 to 34.35] | 9.2 (3.44) [6.25 to 12.14]
  Baseline to 6 month | 34.88 (6.31) [32.02 to 37.74] | 11.60 (6.01) [8.33 to 14.86]
Statistical Analysis 1: Comparison: Mirror Therapy vs Control Group; At Baseline; Test type: Superiority or Other; p = 0.77, t-test, 2 sided; Mean Difference (Final Values) = -0.43, Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: Mirror Therapy vs Control Group; Mean Change from baseline to 1 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 14.12, 95% CI 2-sided [11.02 to 17.25]
Statistical Analysis 3: Comparison: Mirror Therapy vs Control Group; Baseline to 3 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 22.56, 95% CI 2-sided [18.65 to 26.48]
Statistical Analysis 4: Comparison: Mirror Therapy vs Control Group; Baseline to 6 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 23.28, 95% CI 2-sided [18.94 to 27.62]

2. Secondary Outcome: Functional Independence Measure
Description: The FIM consists of 13 motor and 5 social-cognitive items, assessing self-care, sphincter management, transfer, locomotion, communication, social interaction and cognition.14 It uses a 7-level scale anchored by extreme rating of total dependence as 1 and complete independence as 7; the intermediate levels are: 6 modiﬁed independence, 5 supervision or set-up, 4 minimal contact assistance, 3 moderate assistance and 2 maximal assistance.
  For the purpose of analysis we divided FIM into two categories ≤5 dependent, ≥6 independent.
Time Frame: Baseline, 1, 3 and 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Mirror Therapy | Control Group
Number analyzed (Participants) | 27 | 21
participants
  Dependent at Baseline | 27 | 21
  Dependent at 1 month | 26 | 20
  Dependent at 3 months | 18 | 19
  Dependent at 6 months | 15 | 19
Statistical Analysis 1: Comparison: Mirror Therapy vs Control Group; At Baseline; Test type: Superiority or Other; p = 0.99, Chi-squared
Statistical Analysis 2: Comparison: Mirror Therapy vs Control Group; At 1 month; Test type: Superiority or Other; p = 0.99, Chi-squared
Statistical Analysis 3: Comparison: Mirror Therapy vs Control Group; At 3 months; Test type: Superiority or Other; p = 0.03, Chi-squared
Statistical Analysis 4: Comparison: Mirror Therapy vs Control Group; At 6 months; Test type: Superiority or Other; p = 0.004, Chi-squared

3. Primary Outcome: Change From Baseline in Line Bisection Test Scores at 1,3, and 6 Months
Description: The Line Bisection Test (LBT) consisted of three horizontal black lines, 20 cm long, one to the right, one central and one to the left side of a sheet of white paper (21cms X 30 cms). The patients were asked to ﬁnd and mark the centre of each line in turn. Errors away from true midline were measured, with leftward errors being given a negative sign, rightward errors a positive sign.
  We took an absolute value for the change in error. The values for baseline to 1 month were calculated by subtracting baseline values from 1 month values. Then, the mean change was calculated for baseline to 1 month. Similar method was followed for the calculation of mean change in baseline to 3 months and 6 months.
  The patients responses were similar for the three lines that they marked hence we took the first line for the interpretation. None of the patients had extreme errors like missed marking at 3 and 6 months.
Time Frame: Baseline, 1,3 and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cms
Arm/Group | Mirror Therapy | Control Group
Number analyzed (Participants) | 26 | 20
cms
  Baseline | 2.28 [-2.14 to 6.70] | 0.45 [-4.87 to 5.77]
  Baseline to 1 month | 10.42 [7.99 to 12.84] | 4.50 [1.73 to 7.26]
  Baseline to 3 month | 18.26 [14.37 to 22.16] | 9.55 [5.10 to 13.99]
  Baseline to 6 month | 19.03 [15.10 to 22.97] | 10.40 [5.91 to 14.88]
Statistical Analysis 1: Comparison: Mirror Therapy vs Control Group; At Baseline; Test type: Superiority or Other; p = 0.64, t-test, 2 sided; Mean Difference (Final Values) = 1.51, Standard Error of Mean 3.25
Statistical Analysis 2: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 1 month; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = 5.92, 95% CI 2-sided [2.24 to 9.60]
Statistical Analysis 3: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 3 month; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = 8.71, 95% CI 2-sided [2.80 to 14.63]
Statistical Analysis 4: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 6 month; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = 8.63, 95% CI 2-sided [2.67 to 14.60]

4. Primary Outcome: Change From Baseline in Picture Identification Task at 1,3, and 6 Months
Description: PIT consisted of 10 pictures on A4 size paper and patients were asked to identify pictures. More the number of pictures identified, lesser was the neglect.
Time Frame: Baseline, 1,3 and 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pictures
Arm/Group | Mirror Therapy | Control Group
Number analyzed (Participants) | 26 | 20
pictures
  Baseline | 4.84 [4.64 to 5.04] | 4.20 [3.71 to 4.69]
  Baseline to 1 month | 4.88 [4.38 to 5.37] | 1.2 [0.64 to 1.75]
  Baseline to 3 month | 5.16 [4.62 to 5.69] | 1.75 [1.15 to 2.34]
  Baseline to 6 month | 5.16 [4.62 to 5.69] | 1.95 [1.34 to 2.55]
Statistical Analysis 1: Comparison: Mirror Therapy vs Control Group; Baseline; Test type: Superiority or Other; p = 0.99, t-test, 2 sided; Mean Difference (Final Values) = 0.64, Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 1 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.68, 95% CI 2-sided [2.93 to 4.42]
Statistical Analysis 3: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 3 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.41, 95% CI 2-sided [2.61 to 4.21]
Statistical Analysis 4: Comparison: Mirror Therapy vs Control Group; Mean change from baseline to 6 month; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 3.21, 95% CI 2-sided [2.40 to 4.02]

5. Secondary Outcome: Modified Rankin Scale (mRS)
Description: 0 - No symptoms at all / 1 - No significant disability despite symptoms / 2 - Slight disability / 3 -Moderate disability, but able to walk without assistance / 4 - Moderate disability and unable to walk without assistance / 5 - Severe disability / 6 - death
  0-2: Good outcome 3-6: Poor outcome
Time Frame: Baseline, 1,3 and 6 months
Measure: Number; unit: participants
Arm/Group | Mirror Therapy | Control Group
Number analyzed (Participants) | 27 | 21
participants
  Poor outcome at Baseline | 27 | 21
  Poor outcome at 1 month | 25 | 20
  Poor outcome at 3 month | 16 | 19
  Poor outcome at 6 month | 14 | 19
Statistical Analysis 1: Comparison: Mirror Therapy vs Control Group; At Baseline; Test type: Superiority or Other; p = 0.99, Chi-squared
Statistical Analysis 2: Comparison: Mirror Therapy vs Control Group; At month 1; Test type: Superiority or Other; p = 0.99, Chi-squared
Statistical Analysis 3: Comparison: Mirror Therapy vs Control Group; At month 3; Test type: Superiority or Other; p = 0.04, Chi-squared
Statistical Analysis 4: Comparison: Mirror Therapy vs Control Group; At month 6; Test type: Superiority or Other; p = 0.01, Chi-squared

ADVERSE EVENTS:
Arm/Group | Mirror Therapy | Control Group
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/21
Other Adverse Events (participants affected / at risk) | 0/27 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes